CLINICAL TRIAL: NCT04026217
Title: Evaluation of Diaphragmatic Function in Hematological Patients With Acute Hypoxemic Respiratory Failure
Brief Title: Diaphragm Ultrasound as a Powerful Tool in Managing Acute Hypoxemic Respiratory Failure in Hematological Patients
Status: Suspended | Type: Observational
Why Stopped: reduced patients enrolment
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Luigi Vetrugno, Luigi Vetrugno, M.D., Anesthesiology and Intensive Care Clinic, Department of Medicine, University of Udine, Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: 2745
Record Dates: First submitted 2019-06-15; First posted 2019-07-19 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Respiratory Failure; Diaphragm Injury; Ultrasound; Mechanical Ventilation Complication
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute hypoxemic respiratory failure due to parenchymal disfunction is one of the main complications of immunocompromised hematological patients. Mechanical ventilation is frequently needed and diaphragm activity has to be assessed not to worsen ventilator-induced lung injury.

DETAILED DESCRIPTION:
Acute hypoxemic respiratory failure due to parenchymal disfunction is one of the main complications of immunocompromised hematological patients. In these cohort of patients mechanical ventilation is frequently needed in order to restore oxygenation and normocapnia. Since every positive-pressure ventilation regimen may potentially determine pulmonary complications, due to alteration in pressure and volume lung homeostasis and diaphragm activity, also diaphragm function has to be assessed not to worsen ventilator-induced lung injury (VILI). Main targets of VILI are pulmonary interstitium and diaphragm.

Pulmonary interstitium is frequently involved in different mechanism of injury, that derive both from induced tidal volume and positive end expiratory pressure (PEEP). Indeed, large tidal volumes generated during assisted spontaneous breathing may configure non-protective ventilation regimens and the so called "pendelluft phenomenon", that is the intrinsic flow of air within the lung from nondependent to dependent regions without changes in tidal volume, may affect inadequate PEEP values.

Positive-pressure ventilation may also alter diaphragm activity. Recent data show that diaphragm disfunction, considered as an enhanced or reduced thickening fraction, occurs in about 65% of patients undergoing mechanical ventilation.

Since the potential harm of positive-pressure ventilation, the optimization of mechanical ventilation is pivotal to ensure an adequate time-to-recovery without concurring to the onset of further lung and diaphragmatic injury. Neurally Adjusted Ventilatory Assist (NAVA) is a recent modality of mechanical ventilation that delivers ventilatory assistance according to the respiratory effort of the patient, measured by electrical activity of the diaphragm (EAdi). NAVA works proportionally with EAdi values, ensuring a better neuroventilatory efficiency compared to other mechanical ventilation modes and also reducing patient-ventilator asynchrony. According to these features NAVA protocol may be useful in preserving gas exchanges and diaphragm function both in invasive and non-invasive ventilation.

Therefore the evaluation of basal diaphragm activity, the choice of the device for oxygen support administration and the setting of ventilatory parameters may influence hospital stay and outcome of patients affected by acute hypoxemic respiratory failure.

The aim of this study is to evaluate the basal diaphragm activity of acute hypoxemic respiratory failure patients admitted in Intensive Care Unit (ICU) and to record diaphragm activity modifications during the ICU stay in relation to the optimization of medical therapy and, if necessary, according to the need of ventilatory support (invasive or non-invasive ventilation delivered with NAVA protocol).

This study intends to register also daily diaphragm thickening fraction, daily arterial blood gas analysis, failure frequency of non-invasive ventilation, frequency of tracheal intubation, length of mechanical ventilation, length of hospital stay and hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* Hypoxemic respiratory failure in hematological patients (PaO2 < 70 mmHg or P/F < 150)

Exclusion Criteria:

* Patients with positive-pressure ventilation regimen of high flow nasal cannula prior to ICU admission
* Unstable clinical condition (use of vasopressors, acute coronary syndrome...)
* Refusal of treatment or informed consent
* Agitation (RASS ≥+2) or lack of collaboration (Kelly Matthay ≥ 5)
* Multiple organ failure
* Enrollment in other study protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematologic patients with hypoxemic respiratory failure
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Diaphragm thickening fraction | At ICU admission
  Diaphragm thickening fraction measured with echography

SECONDARY OUTCOMES:
Diaphragm thickening fraction | From date of enrollment until the date of death from any cause or ICU discharge, assessed up to 36 months
  Diaphragm thickening fraction measured with echography
Arterial blood gas analysis | From date of enrollment until the date of death from any cause or ICU discharge, assessed up to 36 months
  Arterial blood gas analysis
Failure of non-invasive ventilation | From date of enrollment until the date of death from any cause or ICU discharge, assessed up to 36 months
  Failure of non-invasive ventilation according to hospital NIV protocol
Rate of tracheal intubation | From date of enrollment until the date of death from any cause or ICU discharge, assessed up to 36 months
  Tracheal intubation
Duration of positive-pressure ventilation | From date of enrollment until the date of death from any cause or ICU discharge, assessed up to 36 months
  Duration of positive-pressure ventilation (NIV or mechanical ventilation)
Hospital length of stay | From date of in-hospital admission until the date of hospital discharge, assessed up to 36 months
  Hospital length of stay
In-hospital mortality | From date of in-hospital admission until the date of death from any cause or hospital discharge, assessed up to 36 months
  In-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Vetrugno, Doctor, Principal Investigator — Anesthesiology and Intensive Care Clinic - Department of Medicine - ASUIUD
Locations (1):
- Anesthesiology and Intensive Care Clinic - Department of Medicine - ASUIUD, Udine, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Azoulay E, Thiery G, Chevret S, Moreau D, Darmon M, Bergeron A, Yang K, Meignin V, Ciroldi M, Le Gall JR, Tazi A, Schlemmer B. The prognosis of acute respiratory failure in critically ill cancer patients. Medicine (Baltimore). 2004 Nov;83(6):360-370. doi: 10.1097/01.md.0000145370.63676.fb. PMID 15525848
- [Background] Thiery G, Azoulay E, Darmon M, Ciroldi M, De Miranda S, Levy V, Fieux F, Moreau D, Le Gall JR, Schlemmer B. Outcome of cancer patients considered for intensive care unit admission: a hospital-wide prospective study. J Clin Oncol. 2005 Jul 1;23(19):4406-13. doi: 10.1200/JCO.2005.01.487. PMID 15994150
- [Background] Benoit DD, Vandewoude KH, Decruyenaere JM, Hoste EA, Colardyn FA. Outcome and early prognostic indicators in patients with a hematologic malignancy admitted to the intensive care unit for a life-threatening complication. Crit Care Med. 2003 Jan;31(1):104-12. doi: 10.1097/00003246-200301000-00017. PMID 12545002
- [Background] Boldrini R, Fasano L, Nava S. Noninvasive mechanical ventilation. Curr Opin Crit Care. 2012 Feb;18(1):48-53. doi: 10.1097/MCC.0b013e32834ebd71. PMID 22186215
- [Background] Antonelli M, Conti G, Rocco M, Bufi M, De Blasi RA, Vivino G, Gasparetto A, Meduri GU. A comparison of noninvasive positive-pressure ventilation and conventional mechanical ventilation in patients with acute respiratory failure. N Engl J Med. 1998 Aug 13;339(7):429-35. doi: 10.1056/NEJM199808133390703. PMID 9700176
- [Background] Hess DR. Noninvasive ventilation for acute respiratory failure. Respir Care. 2013 Jun;58(6):950-72. doi: 10.4187/respcare.02319. PMID 23709194
- [Background] Nava S, Hill N. Non-invasive ventilation in acute respiratory failure. Lancet. 2009 Jul 18;374(9685):250-9. doi: 10.1016/S0140-6736(09)60496-7. PMID 19616722
- [Background] Antonelli M, Conti G, Esquinas A, Montini L, Maggiore SM, Bello G, Rocco M, Maviglia R, Pennisi MA, Gonzalez-Diaz G, Meduri GU. A multiple-center survey on the use in clinical practice of noninvasive ventilation as a first-line intervention for acute respiratory distress syndrome. Crit Care Med. 2007 Jan;35(1):18-25. doi: 10.1097/01.CCM.0000251821.44259.F3. PMID 17133177
- [Background] Ferrer M, Esquinas A, Leon M, Gonzalez G, Alarcon A, Torres A. Noninvasive ventilation in severe hypoxemic respiratory failure: a randomized clinical trial. Am J Respir Crit Care Med. 2003 Dec 15;168(12):1438-44. doi: 10.1164/rccm.200301-072OC. Epub 2003 Sep 18. PMID 14500259
- [Background] Agarwal R, Handa A, Aggarwal AN, Gupta D, Behera D. Outcomes of noninvasive ventilation in acute hypoxemic respiratory failure in a respiratory intensive care unit in north India. Respir Care. 2009 Dec;54(12):1679-87. PMID 19961634
- [Background] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464
- [Background] Stephan F, Barrucand B, Petit P, Rezaiguia-Delclaux S, Medard A, Delannoy B, Cosserant B, Flicoteaux G, Imbert A, Pilorge C, Berard L; BiPOP Study Group. High-Flow Nasal Oxygen vs Noninvasive Positive Airway Pressure in Hypoxemic Patients After Cardiothoracic Surgery: A Randomized Clinical Trial. JAMA. 2015 Jun 16;313(23):2331-9. doi: 10.1001/jama.2015.5213. PMID 25980660
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Frat JP, Ragot S, Girault C, Perbet S, Prat G, Boulain T, Demoule A, Ricard JD, Coudroy R, Robert R, Mercat A, Brochard L, Thille AW; REVA network. Effect of non-invasive oxygenation strategies in immunocompromised patients with severe acute respiratory failure: a post-hoc analysis of a randomised trial. Lancet Respir Med. 2016 Aug;4(8):646-652. doi: 10.1016/S2213-2600(16)30093-5. Epub 2016 May 27. PMID 27245914
- [Background] Corley A, Rickard CM, Aitken LM, Johnston A, Barnett A, Fraser JF, Lewis SR, Smith AF. High-flow nasal cannulae for respiratory support in adult intensive care patients. Cochrane Database Syst Rev. 2017 May 30;5(5):CD010172. doi: 10.1002/14651858.CD010172.pub2. PMID 28555461
- [Background] Goligher EC, Dres M, Fan E, Rubenfeld GD, Scales DC, Herridge MS, Vorona S, Sklar MC, Rittayamai N, Lanys A, Murray A, Brace D, Urrea C, Reid WD, Tomlinson G, Slutsky AS, Kavanagh BP, Brochard LJ, Ferguson ND. Mechanical Ventilation-induced Diaphragm Atrophy Strongly Impacts Clinical Outcomes. Am J Respir Crit Care Med. 2018 Jan 15;197(2):204-213. doi: 10.1164/rccm.201703-0536OC. PMID 28930478
- [Background] Wait JL, Nahormek PA, Yost WT, Rochester DP. Diaphragmatic thickness-lung volume relationship in vivo. J Appl Physiol (1985). 1989 Oct;67(4):1560-8. doi: 10.1152/jappl.1989.67.4.1560. PMID 2676955
- [Background] Cohn D, Benditt JO, Eveloff S, McCool FD. Diaphragm thickening during inspiration. J Appl Physiol (1985). 1997 Jul;83(1):291-6. doi: 10.1152/jappl.1997.83.1.291. PMID 9216975
- [Background] Goligher EC, Ferguson ND, Brochard LJ. Clinical challenges in mechanical ventilation. Lancet. 2016 Apr 30;387(10030):1856-66. doi: 10.1016/S0140-6736(16)30176-3. Epub 2016 Apr 28. PMID 27203509
- [Background] Contejean A, Lemiale V, Resche-Rigon M, Mokart D, Pene F, Kouatchet A, Mayaux J, Vincent F, Nyunga M, Bruneel F, Rabbat A, Perez P, Meert AP, Benoit D, Hamidfar R, Darmon M, Jourdain M, Renault A, Schlemmer B, Azoulay E. Increased mortality in hematological malignancy patients with acute respiratory failure from undetermined etiology: a Groupe de Recherche en Reanimation Respiratoire en Onco-Hematologique (Grrr-OH) study. Ann Intensive Care. 2016 Dec;6(1):102. doi: 10.1186/s13613-016-0202-0. Epub 2016 Oct 25. PMID 27783381
- [Background] Talmor D, Sarge T, Malhotra A, O'Donnell CR, Ritz R, Lisbon A, Novack V, Loring SH. Mechanical ventilation guided by esophageal pressure in acute lung injury. N Engl J Med. 2008 Nov 13;359(20):2095-104. doi: 10.1056/NEJMoa0708638. Epub 2008 Nov 11. PMID 19001507
- [Background] Brochard L, Slutsky A, Pesenti A. Mechanical Ventilation to Minimize Progression of Lung Injury in Acute Respiratory Failure. Am J Respir Crit Care Med. 2017 Feb 15;195(4):438-442. doi: 10.1164/rccm.201605-1081CP. PMID 27626833
- [Background] Carteaux G, Millan-Guilarte T, De Prost N, Razazi K, Abid S, Thille AW, Schortgen F, Brochard L, Brun-Buisson C, Mekontso Dessap A. Failure of Noninvasive Ventilation for De Novo Acute Hypoxemic Respiratory Failure: Role of Tidal Volume. Crit Care Med. 2016 Feb;44(2):282-90. doi: 10.1097/CCM.0000000000001379. PMID 26584191
- [Background] L'Her E, Deye N, Lellouche F, Taille S, Demoule A, Fraticelli A, Mancebo J, Brochard L. Physiologic effects of noninvasive ventilation during acute lung injury. Am J Respir Crit Care Med. 2005 Nov 1;172(9):1112-8. doi: 10.1164/rccm.200402-226OC. Epub 2005 Aug 4. PMID 16081548
- [Background] Mauri T, Cambiaghi B, Spinelli E, Langer T, Grasselli G. Spontaneous breathing: a double-edged sword to handle with care. Ann Transl Med. 2017 Jul;5(14):292. doi: 10.21037/atm.2017.06.55. PMID 28828367
- [Background] Goligher EC, Kavanagh BP, Rubenfeld GD, Adhikari NK, Pinto R, Fan E, Brochard LJ, Granton JT, Mercat A, Marie Richard JC, Chretien JM, Jones GL, Cook DJ, Stewart TE, Slutsky AS, Meade MO, Ferguson ND. Oxygenation response to positive end-expiratory pressure predicts mortality in acute respiratory distress syndrome. A secondary analysis of the LOVS and ExPress trials. Am J Respir Crit Care Med. 2014 Jul 1;190(1):70-6. doi: 10.1164/rccm.201404-0688OC. PMID 24919111
- [Background] Stenqvist O, Grivans C, Andersson B, Lundin S. Lung elastance and transpulmonary pressure can be determined without using oesophageal pressure measurements. Acta Anaesthesiol Scand. 2012 Jul;56(6):738-47. doi: 10.1111/j.1399-6576.2012.02696.x. Epub 2012 Apr 23. PMID 22524531
- [Background] Hedenstierna G. Esophageal pressure: benefit and limitations. Minerva Anestesiol. 2012 Aug;78(8):959-66. Epub 2012 Jun 14. PMID 22699701
- [Background] Terzi N, Piquilloud L, Roze H, Mercat A, Lofaso F, Delisle S, Jolliet P, Sottiaux T, Tassaux D, Roesler J, Demoule A, Jaber S, Mancebo J, Brochard L, Richard JC. Clinical review: Update on neurally adjusted ventilatory assist--report of a round-table conference. Crit Care. 2012 Jun 20;16(3):225. doi: 10.1186/cc11297. PMID 22715815
- [Background] Colombo D, Cammarota G, Bergamaschi V, De Lucia M, Corte FD, Navalesi P. Physiologic response to varying levels of pressure support and neurally adjusted ventilatory assist in patients with acute respiratory failure. Intensive Care Med. 2008 Nov;34(11):2010-8. doi: 10.1007/s00134-008-1208-3. Epub 2008 Jul 16. PMID 18629471
- [Background] Schmidt M, Kindler F, Cecchini J, Poitou T, Morawiec E, Persichini R, Similowski T, Demoule A. Neurally adjusted ventilatory assist and proportional assist ventilation both improve patient-ventilator interaction. Crit Care. 2015 Feb 25;19(1):56. doi: 10.1186/s13054-015-0763-6. PMID 25879592
- [Background] Di Mussi R, Spadaro S, Mirabella L, Volta CA, Serio G, Staffieri F, Dambrosio M, Cinnella G, Bruno F, Grasso S. Impact of prolonged assisted ventilation on diaphragmatic efficiency: NAVA versus PSV. Crit Care. 2016 Jan 5;20:1. doi: 10.1186/s13054-015-1178-0. PMID 26728475

DOCUMENTS (2):
  • Study Protocol (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT04026217/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT04026217/SAP_001.pdf